CLINICAL TRIAL: NCT06940700
Title: To Evaluate the Efficacy and Safety of SHR-4597 Inhalants in Adults With Asthma: a Multicenter, Randomized, Open-label, Positive-controlled Phase II Clinical Study
Brief Title: Clinical Study on the Efficacy and Safety of SHR-4597 Inhalant in Adult Patients With Asthma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-4597-201
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A (Experimental): SHR4597
  Interventions: Drug: SHR4597
- Treatment group B (Experimental): SHR4597
  Interventions: Drug: SHR4597
- Treatment group C (Active Comparator): Budesonide inhalant
  Interventions: Drug: Budesonide inhalant

INTERVENTIONS:
Drug: SHR4597 — SHR4597
  Arms: Treatment group A; Treatment group B
Drug: Budesonide inhalant — Budesonide inhalant
  Arms: Treatment group C

SUMMARY:
To evaluate the efficacy and safety of SHR-4597 inhalants in adults with asthma: a multicenter, randomized, open-label, positive-controlled Phase II clinical study

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old and ≤75 years old, gender is not limited;
2. Body mass index (BMI) ≥18 and ≤30 kg/m2 during screening period;
3. Medical history and objective evidence consistent with current guidelines supporting an asthma diagnosis within the 12 months prior to randomization;
4. Did not receive inhaled corticosteroids (ICS) and/or combined with other asthma control medications within 2 weeks prior to randomization;
5. FEV1 during the screening period and before bronchodilator inhalation at baseline accounted for ≥40% and < 80% of the estimated value;
6. Screening and baseline visit, Asthma Control Questionnaire-6 (ACQ-6) score ≥1.5;
7. FeNO values at screening period and baseline ≥25 ppb;
8. Patients with asthma who were treated for the first time or who had previously taken irregular medication were selected; Among them, the definition of irregular past use was: patients did not regularly use asthma control drugs within the first 3 months of enrollment, and the average weekly use compliance was < 50%.
9. A fertile female subject or a male subject whose partner is a fertile female must agree not to have a family plan and to voluntarily use highly effective contraception (including the partner) from the time of signing the informed consent until 1 month after the last study drug administration, and refrain from sperm/egg donation;
10. Voluntarily sign informed consent to participate in this study.
11. The subjects were unable to complete the questionnaires due to their limited educational level, or neither the subjects themselves nor their families could fill in the subject log card.
12. The researchers determined that there were other circumstances that were not suitable for participation in this study.

Exclusion Criteria:

1. Combined diseases or conditions

   * Clinically significant pulmonary diseases, including but not limited to active pulmonary tuberculosis, bronchiectasis, atelectasis, idiopathic pulmonary fibrosis, bronchopulmonary aspergillosis, and chronic obstructive pulmonary disease (COPD);

     * Malignant tumors diagnosed within 5 years prior to randomization (except those with a low risk of metastasis and death, such as well-treated basal cell carcinoma of the skin or carcinoma in situ of the cervix);

       * Combined with poorly controlled hypertension (systolic blood pressure ≥180mmHg, and/or diastolic blood pressure ≥110mmHg during the screening period) or uncontrolled severe cardiovascular and cerebrovascular diseases; ④ Known immunodeficiency;

         * A history of infection requiring clinical intervention within 4 weeks prior to randomization, including but not limited to respiratory infection;

           ⑥ Known presence of parasitic infection within 6 months prior to randomization;

           ⑦ Blood donation or significant blood loss (≥400ml), or transfusion of blood products or immunoglobulin within 4 weeks prior to randomization;

           ⑧ A history of life-threatening acute asthma attacks (including admission to the intensive care unit and/or the need for invasive ventilator support [intubation/tracheotomy]);

           ⑨ History of acute asthma attack in the 4 weeks prior to randomization.
2. Combination of medication or treatment

   * Receiving non-selective beta-blockers (e.g., propranolol) within 1 week prior to screening;

     * Live attenuated vaccine or recombinant vaccine with viral vector were received within 4 weeks before randomization;

       * Receiving allergen immunotherapy 8 weeks before randomization;

         * Within 12 weeks before randomization or within 5 half-lives of the drug (refer to the drug instructions, whichever is older; For those with unknown half-lives, the first 12 weeks of randomization will be the use of systemic immunosuppressants (except for systemic glucocorticoids for asthma treatment, and systemic glucocorticoids for other conditions <3 days) or immunomodulators, or biologics or Th2 cytokine inhibitors, Including but not limited to methotrexate, cyclosporine, interferon-alpha, anti-IL-5 monoclonal antibody,anti-TSLP monoclonal antibody, anti-IGE monoclonal antibody, mesulast, etc.

           * Receiving a single dose of long-acting β2 agonist within 4 weeks prior to screening; ⑥4 weeks before randomization, inhaled corticosteroids (>500 micrograms of beclomethasone dipropionate per day [BDP] or equivalent dose);

             ⑦4 weeks before randomization, systemic glucocorticoid therapy;
             * Received bronchial thermoplasty or bronchial cryoablation within 1 year before randomization; ⑨There is a surgical plan during the study, or other treatment that the investigator believes may affect the evaluation of the subject;
3. Laboratory examination

   ①Significant abnormalities during screening or baseline laboratory tests:
   1. White blood cell (WBC) < 3.0×109/L;
   2. Blood eosinophils >1500cells/μL (1.5×109/L)
   3. Hemoglobin (Hb) ≤90 g/L;
   4. Alanine aminotransferase (ALT) > 3×ULN (upper limit of normal);
   5. Aspartate aminotransferase (AST) > 3×ULN;
   6. Total bilirubin (TBIL) > 1.5×ULN;
   7. Prothrombin time (PT) > ULN+3s;
   8. Creatinine (Cr) > 1.5×ULN;
   9. Co-active hepatitis B (peripheral blood hepatitis B virus deoxyribonucleic acid (HBV DNA) ≥1×103 IU[or copy] / mL), or hepatitis C antibody positive, or human immunodeficiency virus (HIV) positive, or treponema pallidum antibody positive.

      * Prolonged ECG QTc interval (>450ms) or other clinically significant abnormal results that may pose significant safety risks to subjects during the screening period;
4. General situation

   * Smoking or smoking cessation less than 6 months during the screening period, or previous smoking ≥10 pack years (pack years = number of years of smoking × number of packs per day); ②A history of drug use, alcohol abuse (average weekly consumption of ≥14 units of alcohol: 1 unit = 285 mL for beer, 25 mL for spirits, or 100 ml for wine) or drug abuse in the year prior to screening;

     * Have participated in other clinical studies and used investigational drugs containing active ingredients within 30 days prior to screening, or have been within 5 half-lives of investigational drugs at the time of screening (whichever is older);

       * Subjects who are pregnant (screening or baseline blood pregnancy test positive) or who plan to become pregnant while breastfeeding or during the study; ⑥Other reasons deemed unsuitable for study participation by the researcher.
       * Excessive alcohol consumption and drug abuse were prohibited throughout the study period (the definition of excessive alcohol consumption is the same as exclusion criterion IV.2).

         * Smoking (including e-cigarettes) was prohibited throughout the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in FEV1 (Pre-BD) from baseline | 6 weeks

SECONDARY OUTCOMES:
Changes in FEV1 before bronchodilator (Pre-BD) administration compared with baseline at week 42 | at week 42
Changes in forced vital capacity (FVC) before bronchodilator (Pre-BD) use compared with baseline at week 42 | at week 42
Changes in peak expiratory flow (PEF) before bronchodilator (Pre-BD) use compared with baseline at week 42 | at week 42
Changes in exhaled nitric oxide (FeNO) from baseline at 42 weeks | at 42 weeks
Changes in Asthma Control Questionnaire (ACQ-6) scores from baseline at 42 weeks | at 42 weeks
Change in mean number of nightly awakenings from baseline over 42 weeks | 42 weeks
Changes in ACT questionnaire scores from baseline at 42 weeks | at 42 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided